CLINICAL TRIAL: NCT04032522
Title: Neonatal HIV Early Infant Diagnosis (EID) Versus Standard of Care EID - Long Term Impact on inFant hEalth: a Feasibility Study of point-of Care Testing at Birth Versus at 6 Weeks of Age, on the Uptake of ART and Infant Prophylaxis, and on Rates of Infant Survival, Morbidity and Retention in Care
Brief Title: Neonatal HIV Early Infant Diagnosis (EID) Versus Standard of Care EID- Long Term Impact on inFant hEalth (LIFE)
Acronym: LIFE
Status: Completed | Type: Observational
Sponsor: Michael Hoelscher (Other)
Collaborators: Instituto Nacional de Saúde, Mozambique (Other Government); NIMR- Mbeya Medical Research Centre (MMRC), Mbeya, Tanzania (Unknown); University of Lisbon Instituto Universitário Egas Moniz (IUEM) Lisbon, Portugal (Unknown); Clinton Health Access Initiative Inc. (Other)
Responsible Party: Sponsor-Investigator, Michael Hoelscher, Director, Division of Infectious Diseases and Tropical Medicine, University Hospital, LMU Munich, Ludwig-Maximilians - University of Munich
Organization: Ludwig-Maximilians - University of Munich (Other)
Other Study IDs: LMU-IMPH-LIFE
Record Dates: First submitted 2019-07-23; First posted 2019-07-25 (Actual); Last update posted 2024-08-22 (Actual); Status verified 2024-08

CONDITIONS: HIV, Neonatal HIV Early-Infant-Diagnosis (EID), Point-of-Care Testing (PoC)
MeSH Terms: interventions — Point-of-Care Systems

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Intervention Arm (A): Half of the health facilities will implement the intervention package. All mothers will be tested using PoC-VL at delivery and all HIV-exposed infants will be offered PoC-EID at birth and week 4-8. Newborns found to be HIV-positive will be offered immediate ART. Neonatal ART initiation will be supported at birth by trained nurses/midwives, and approved and supervised by local doctors from the affiliated HIV CTC. Following ART initiation infants will be referred for consolidated ART management to their paediatric HIV clinic following local procedures. Newborns testing HIV-negative will be offered postnatal prophylaxis (PNP) or enhanced postnatal prophylaxis (ePNP), depending on clinical risk factors, the maternal VL and country guidelines. Mothers with HIV-RNA >1000 copies/mL will receive immediate referral information for ART initiation if not on ART or enhanced ART counselling, with follow up virologic testing and switch of ART regimen as applicable at their local HIV clinic.
  Interventions: Other: point-of care (PoC) neonatal HIV early infant diagnosis (EID)
- Control Arm (B): The other half of the health facilities will implement the standard of care (SoC). Enrolled mothers will not receive immediate PoC VL at delivery, but infants deemed to be at high risk using clinical criteria (e.g. no or late initiation of maternal ART) will be offered ePNP. EID testing will follow the national algorithm with testing at 4-8 weeks, followed by referral for immediate ART initiation for all HIV-infected infants. As PoC EID testing is expected to be nationally implemented on a programme level we will facilitate the availability of PoC testing at these sites.

INTERVENTIONS:
Other: point-of care (PoC) neonatal HIV early infant diagnosis (EID) — clinical impact of a PoC-EID for infants and neonates at birth and week 4-8 weeks, linked with nurse-supported immediate ART initiation in HIV-infected neonates, versus standard-of-care (SoC)
  Groups: Intervention Arm (A)

SUMMARY:
This study we will evaluate the benefit of HIV testing in neonates born from HIV-infected mothers in Tanzania and Mozambique. The study will use and evaluate novel point-of-care diagnostic systems, that can provide neonatal HIV test results within 2 hours. We will evaluate if HIV testing at birth followed by immediate neonatal HIV treatment initiation will lead to lesser infant's sickness, HIV progression or even death as compared to the current standard procedure which is infant HIV testing at week 6 after delivery. This will be associated with a cost-effectiveness analysis in order to guide national HIV programs for their guidelines. The study will further evaluate if point-of care viral load testing in mothers at birth will identify high-risk scenarios for HIV transmission from the mother to her child. This should lead to enhanced prophylactic treatments in HIV-exposed infants and we hypothesize that PoC VL monitoring at birth leads to lower transmission rates. The study will be performed at 28 maternity health facilities in Tanzania and Mozambique, half of them will be randomized to provide birth HIV PoC infant and maternal viral load testing, the other half will provide the current standard of care (infant HIV testing at week 6, no PoC VL monitoring at birth for the mother). The study is conducted in public health settings, and some study objectives also focus on how successful modern HIV treatments can be provided to infants, if HIV testing and treatment procedures are feasible for nurses and midwives, and if these procedures can be carried out in a timely manner. This study also includes a basic research component that will investigate how HIV spreads in the body of HIV-infected infants, and if early infant HIV diagnosis and treatment can reduce the spread in cells of HIV-infected individuals.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntary and informed consent of the mother for her own study participation
2. Voluntary and informed consent of the legal guardian of the child for participation of the child in the study.
3. Mothers/legal guardians ≥18 years of age.
4. Documented maternal HIV infection.
5. Willingness to consent to HIV testing for the child and herself.
6. Willingness to consent to active tracing including home tracing.

Exclusion Criteria:

1. Deficiency in the mother, rendering it difficult, if not impossible, for her or her infant to take part in the study or understand the information provided to her. This includes alcoholism, drug dependency as well as psychiatric illnesses, suicidal tendencies or any other inability.
2. Having delivered more than 72h (3 days) ago
3. Prisoners
4. Women presenting with an emergency requiring immediate medical assistance if not resolved at study inclusion
5. Stillbirths
6. Infant requiring emergency care (e.g. immediate or rapid occurring life threatening conditions, resuscitation, prolonged obstetric related intensive care, severe jaundice) or born with severe malformation.
7. If within the discretion of the investigator based on recommendation of the gynaecologist or paediatrician in charge study participation would possibly add not acceptable risk or burden to the mother or infant (e.g. significant congenital malformation, health deficiencies, very low birth weight less than 1500g)
8. Unlikely to comply with protocol as judged by the principal investigator or his designate

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: HIV infected pregnant women and their exposed infants will be recruited at maternity clinics in Mozambique and Tanzania. Assuming a 4% MTCT rate by week 6 and a difference of combined HIV-infected infant endpoints of 14% (Arm A) versus 30% (Arm B) the study target is to enrol at least 224 HIV infected infants (112 per arm) from both countries into the follow-up phase resulting in an overall recruitment number of 6000 mother-child pairs (3000 per arm), including an assumed 5% loss to follow-up. Furthermore, we will enrol 400 HIV-exposed infants from both countries after week 12 into a long-term follow-up phase to investigate MTCT rates and associated MTCT risks until the end of the study period after cessation of breastfeeding.
Sampling Method: Probability Sample
Enrollment: 6602 (Actual)
Dates: Start 2019-10-23 (Actual); Primary Completion 2023-01-01 (Actual); Study Completion 2023-01-01 (Actual)

PRIMARY OUTCOMES:
clinical impact of a PoC-EID | Proportion of combined clinical endpoints in HIV-infected infants at months 18 between arms
  The primary objective is to establish the clinical impact of a PoC-EID for infants and neonates at birth and week 4-8 weeks, linked with nurse-supported immediate ART initiation in HIV-infected neonates, versus standard-of-care (SoC) on the primary and secondary endpoints. Combined clinical outcomes will include mortality, morbidity (WHO Stage 2 or above disease, severe infant medical conditions), hospitalization, toxicity (Grade 3 or above laboratory abnormality), poor antiretroviral treatment response (confirmed virological failure, treatment termination or prolonged interruption), or loss to follow up of HIVinfected infants.

CONTACTS AND LOCATIONS:
Overall Officials: Arne Kroidl, Dr. med, Study Chair — Division of Infectious Diseases and Tropical Medicine, University Hospital, LMU Munich; Ilesh Jani, Dr., Ph.D., Principal Investigator — Instituto Nacional de Saúde, Mozambique; Issa Sabi, Dr., Principal Investigator — NIMR- Mbeya Medical Research Centre (MMRC), Mbeya, Tanzania
Locations (2):
- Centro de Investigacao Operacional da Beira (CIOB), Beira, Sofala, Mozambique
- Mbeya Medical Research Centre, Mbeya, Tanzania

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Jani IV, Sabi I, Elsbernd K, Meggi B, Mahumane A, Lwilla AF, Pereira K, Boniface S, Edom R, Lequechane J, Chale F, Chiwerengo N, Ntinginya NE, Mudenyanga C, Mueller M, Rauscher M, Hoelscher M, Taveira N, Buck WC, Kroidl A; LIFE Study Consortium. Impact of Point-of-Care Birth Test-and-Treat on Clinical Outcomes Among Infants With HIV: A Cluster-Randomized Trial in Mozambique and Tanzania. Clin Infect Dis. 2025 Jun 4;80(5):1114-1124. doi: 10.1093/cid/ciae530. PMID 39514367